CLINICAL TRIAL: NCT02381392
Title: A Comparison of Accuvein to Standard Intravenous Access in Children 0 to 24 Months of Age in the Pediatric Emergency Department
Brief Title: A Comparison of Accuvein to Standard IV Access in Children 0 to 24 Months of Age in the Pediatric ED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment, investigator left institution
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Kelly Young, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21283-01
Record Dates: First submitted 2015-02-21; First posted 2015-03-06 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Disorder
Keywords: emergency medicine; infrared; intravenous

STUDY DESIGN:
Intervention Model Description: Intervention group using Accuvein, Control group standard care
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AV400 (Experimental): The nurse will use the Accuvein AV400 to assist with intravenous access. If the nurse cannot place the catheter after 2 tries (two needle sticks into the skin) then the nurse will attempt to put in the catheter without using the device. While the nurse is putting in the catheter, a member of the study team will record the number of tries, the type of catheter and where the catheter is successfully put in. Afterwards the parent and nurse will be surveyed on their satisfaction and the nurse will be asked specific questions about using the AV400.
  Interventions: Device: Accuvein AV400
- Standard (No Intervention): The nurse will use the standard technique for intravenous access (not using the Accuvein AV400). If the nurse cannot place the catheter after 2 tries (two needle sticks into the skin) then the nurse will attempt to put in the catheter with the help of the Accuvein AV400. While the nurse is putting in the catheter, a member of the study team will record the number of tries, the type of catheter and where the catheter is successfully put in. Afterwards the parent and nurse will be surveyed on their satisfaction and the nurse will be asked specific questions about using the AV400 if they crossed over to the AV400 after two failures.

INTERVENTIONS:
Device: Accuvein AV400 — This device is FDA approved for assistance with intravenous access. It has been shown to cause no harm to patients. The device utilizes infrared technology to provide a visible map of the subject's blood vessels where the light is shone.
  Arms: AV400

SUMMARY:
Obtaining intravenous (IV) access in children under the age of 2 years is difficult, especially in the emergency department (ED) where the children can be frightened, dehydrated and ill. Often it requires multiple needle sticks and nurses to place an IV in a difficult child. In our ED the recently acquired an Accuvein AV400 device. This infrared light, like a barcode scanner, makes the veins on a child appear like roads on a map. This ideally shows the nurse where to place and direct the needle. This device is approved by the FDA to work with children and has not been shown to have any harmful effects. However, there are no studies showing whether this device helps in the difficult less than 2 year olds seen in the emergency department.

This study will be to directly compare placing an IV in a child under 2 years of age with the AV400 versus not using the device. A physician, medical student, or nurse practitioner who has been trained on how to observe nurses place IVs will enroll children who require an IV for their ED clinical care (as determined by their ED doctors). This person will consent the parents, ask the parents questions regarding the child's past medical history, and have the nurse look at the veins of the child ahead of the IV access attempt to rate the level of difficulty expected (easy, moderate, difficult). Whether the child has the IV attempt performed with or without the AV400 will be computer randomized. The nurse will attempt to place the IV, and the study staff will observe and record the number of attempts, size of the IV catheter, and location of the IV. If 2 attempts are failed, the patient will "cross over" to the other condition, that is if AV400 was being used then it will not be used, and if AV400 was not being used then it will be used. If there are 4 failed attempts at IV placement, then the child will be treated as per our department's difficult IV access protocol, which is applied to all children with difficult IV access regardless of participation in the study. After the IV placement, both the parents and the nurse will be asked several questions regarding satisfaction with use of the AV400.

No patient identifiers will be collected.

The investigators will be recruiting 260 children to determine if using the AV400 device improves the first time needle stick success from 40% to 60%.

Nursing approval for the study was obtained prior to the study.

DETAILED DESCRIPTION:
The investigators hypothesize that the use of the Accuvein AV400 (AV400) with intravenous access will improve the first attempt success rate in intravenous (IV) starts for patients ages 0-24 months of age by 20% as compared to the standard technique.

Study Recruitment and protocol

* Potential subjects will be patients age 0-24 months recruited from the pediatric emergency department at Harbor-UCLA. The patients will be screened for meeting criteria of age 0-24 months, requiring IV access, not requiring emergent resuscitative access, and not being a ward of the state.
* Nurses who work in the pediatric emergency department and who obtain IV access in children will be solicited by members of the research team to participate in the study. All nurses who are trained to use the device will be able to participate as operators in the study.
* The patient will be enrolled as a subject and the data collection form will be filled out by a trained observer. The data collection form contains: trained observer level of training; blinded nursing number; randomization number; patient gender, age in months, weight, height, Fitzpatrick skin color, dehydration status, mental status, gestational age, chronic medical conditions, and hospitalizations in last two years; nurse's assessment of vein palpability, visibility, and subjective difficulty; nurse's pediatric ED experience and overall experience in years; access tool and whether crossover was utilized; IV gauge, IV access site, number of persons needed to assist, and whether access was successful. All trained observers will have undergone training to ensure reliability between observers. Once a patient has been identified as a potential subject by the trained observer and consent has been obtained, a blinded randomized manila envelope will be chosen. The data collection form will be completed by the trained observer and then the nurse will attempt first IV attempt per the arm of the study (standard versus with AV400 assistance). The patient will receive two attempts using the assigned randomized method. If 2 failed attempts, the nurse will cross arms of the study and use the other IV access method. If this fails, the standard difficult IV access pathway used by the pediatric ED will be started. Currently this pathway is started after 4 failed IV attempts. Therefore, there is no additional risk to the subject in the study. After the IV access has been successful or the difficult IV access pathway has begun, the trained observer will then ask the parent and nurse a series of questions based on a Likert scale to assess satisfaction and whether the nurse felt the AV400 helped find veins, distracted her/him from usual technique, and/or saved time. No identifying data will be collected on the nurse or subject. Trained observers will not be ordering any IV placements, labs or medications for subjects. Potential subjects will have had orders placed for IV access prior to their selection for eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric emergency department patient age 0-24 months who requires intravenous access. Patients requiring emergent resuscitation will not be included.

Exclusion Criteria:

* Treatment will not be delayed to consent the patient's parent. If consent cannot be obtained by the study team in a timely manner, the patient will not be eligible to be included in the study.
* Subjects who are in foster care or in the care of the state.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11-19 (Actual); Study Completion 2016-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Young, MD, MS, Principal Investigator — Harbor-UCLA Department of Emergency Medicine; Joelle Donofrio, DO, Study Director — Harbor-UCLA Department of Emergency Medicine
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AV400 | Standard
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AV400 | Standard | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 12 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23
Fitzpatrick skin color [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color. Patients are graded as follows:
  Type I always burns, never tans (pale white; blond / red hair; blue eyes; freckles).
  Type II usually burns, tans minimally (white; fair; blond / red hair; blue, green, or hazel eyes) Type III sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV burns minimally, always tans well (moderate brown) Type V very rarely burns, tans very easily (dark brown)
  Participants
    I | 0 | 0 | 0
    II | 4 | 2 | 6
    III | 5 | 8 | 13
    IV | 1 | 2 | 3
    V | 1 | 0 | 1
Dehydration status [Count of Participants; unit: Participants]
  None | 2 | 4 | 6
  Mild | 9 | 5 | 14
  Moderate | 0 | 1 | 1
  Missing data | 0 | 2 | 2
Mental status [Count of Participants; unit: Participants]
  Combative | 7 | 8 | 15
  Cooperative | 3 | 3 | 6
  Missing data | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success at Intravenous Access
Description: Successful: Intravenous line successfully placed with blood able to be drawn back and fluid able to be flushed into the vein. Flashback but IV blown: blood initially successfully drawn back or seen in the syringe, but subsequently unable to flush fluid into the vein. No flashback: no blood drawn back into or seen in the syringe at all. Missing data: data not recorded regarding success or flashback.
Time Frame: Intravenous access attempts during the current emergency department visit only, average of 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AV400 | Standard
Number analyzed (Participants) | 11 | 12
Participants
  Successful | 3 | 7
  Flashback but IV blown | 5 | 3
  No flashback | 2 | 2
  Missing data | 1 | 0

2. Secondary Outcome: Median Number of Intravenous Attempts
Description: To compare the median number of IV access attempts until success or escalation of therapy to the difficult IV access team between those placed with the AV400 as to those without (ie the standard technique).
Time Frame: Intravenous access attempts during the current emergency department visit only, average of 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AV400 | Standard
Number analyzed (Participants) | 11 | 12
Participants
  1 | 3 | 7
  2 | 4 | 3
  3 | 1 | 2
  5 or more | 2 | 0
  Missing data | 1 | 0

3. Secondary Outcome: Parent Satisfaction (Likert Scale)
Description: To compare parent satisfaction using a Likert scale between use of the AV400 and the standard technique
Time Frame: Intravenous access attempts during the current emergency department visit only, average of 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AV400 | Standard
Number analyzed (Participants) | 11 | 12
Participants
  Extremely satisfied | 0 | 3
  Very satisfied | 0 | 2
  Satisfied | 2 | 2
  Partially satisfied | 6 | 3
  Dissatisfied | 1 | 0
  Missing data | 2 | 2

4. Secondary Outcome: Nursing Satisfaction (Likert Scale)
Description: To compare nursing satisfaction using a Likert scale between use of the AV400 and the standard technique.
Time Frame: Intravenous access attempts during the current emergency department visit only, average of 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AV400 | Standard
Number analyzed (Participants) | 11 | 12
Participants
  Extremely satisfied | 0 | 1
  Very satisfied | 3 | 1
  Satisfied | 2 | 5
  Partially satisfied | 3 | 1
  Dissatisfied | 1 | 2
  Missing data | 2 | 2

5. Secondary Outcome: Success in Patients With High Difficult Intravenous Access Scores
Description: as for outcome 1
Time Frame: Intravenous access attempts during the current emergency department visit only, average of 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | AV400 | Standard
Number analyzed (Participants) | 4 | 5
Participants
  Successful | 2 | 4
  Flashback but IV blown | 1 | 0
  No flashback | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events collected only during participation in the study (during the emergency department visit only), for an average duration of 120 minutes
Description: No difference
Arm/Group | AV400 | Standard
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

LIMITATIONS AND CAVEATS:
Unable to complete enrollment in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No